CLINICAL TRIAL: NCT00232674
Title: The Effect of Inhaled Corticosteroids on the Development of Emphysema in Smokers Assessed by Computed Tomography (CT).
Brief Title: Efficacy Study of the Effect of Budesonide on Emphysema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-004-0001
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

INTERVENTIONS:
Drug: Pulmicort (budesonide) Turbuhaler

SUMMARY:
To assess the effect of up to 4 years treatment with budesonide on progression of emphysema in patients with Chronic Obstructive Lung Disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Chronic Obstructive Pulmonary Disease diagnosis
* smoker

Exclusion Criteria:

* No exacerbation within the last 30 days
* no long term use of oral corticosteroids

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 1999-07; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
The primary variable in the study was change in lung density measured by Computed Tomography annually.

SECONDARY OUTCOMES:
Decline in lung Function (FEV1) and exacerbation rate were measured biannually and decline in diffusion capacity (TLCO) annually.

CONTACTS AND LOCATIONS:
Overall Officials: Astra Zeneca, Study Director — AstraZeneca
Locations (1):
- Research Site, Gentofte Municipality, Denmark